CLINICAL TRIAL: NCT01273714
Title: Subtotal Versus Total Thyroidectomy for Benign Thyroid Disease - a Prospective Case-control Surgical Outcome Study.
Brief Title: Subtotal Versus Total Thyroidectomy for Benign Goiter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BBN/501/ZKL/87/L
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Goiter
Keywords: benign thyroid disease; incidental thyroid cancer; recurrent goiter; revision thyroid surgery
MeSH Terms: conditions — Goiter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BST (Active Comparator): bilateral subtotal thyroidectomy (leaving on both sides of the neck thyroid stumps of approximately 2 g of normal remnant tissue each)
  Interventions: Procedure: thyroid resection
- TT (Experimental): extracapsular total thyroidectomy
  Interventions: Procedure: thyroid resection

INTERVENTIONS:
Procedure: thyroid resection — bilateral subtotal versus total thyroidectomy

SUMMARY:
The extent of thyroid resection in benign goiter is controversial. Potential advantages of TT over BST may include: one-stage removal of incidental thyroid cancer reported in up to 10% of operatively treated benign thyroid diseases, and lower risk for goiter recurrence. However, these potential advantages should outweigh the risk of morbidity associated with more radical thyroid resection.

The aim of this study was to compare outcomes of bilateral subtotal (BST) vs. total thyroidectomy (TT) for benign bilateral thyroid disease.

DETAILED DESCRIPTION:
The extent of thyroid resection in bilateral multinodular non-toxic goiter remains controversial. Surgeons still continue to debate whether the potential benefits of total thyroidectomy outweigh the potential complications. Most low-volume surgeons avoid to perform total thyroidectomy owing to the possible complications such as permanent recurrent laryngeal nerve palsy and permanent hypoparathyroidism. On the other hand, the increasing number of total thyroidectomies are currently performed in high-volume endocrine surgery units, and the indication for this procedure include thyroid cancer, Graves disease and multinodular goiter. Recently there has been increasing acceptance for performing total thyroidectomy for bilateral multinodular non-toxic goiter as it removes the disease process completely, lowers local recurrence rate and avoids the substantial risk of reoperative surgery, and involves only a minimal risk of morbidity. This common perception is based largely on single-institution retrospective data, a few multi-institutional retrospective experiences, and only a few small prospective studies comparing the outcomes of total vs. subtotal thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* a benign bilateral thyroid disease with the posterior aspects of both thyroid lobes appearing normal on ultrasound of the neck.

Exclusion Criteria:

* thyroid disease involving the posterior aspect/s of thyroid lobe/s,
* suspicion of thyroid cancer,
* previous thyroid surgery,
* pregnancy or lactation,
* age < 18 years or > 65 years,
* ASA 4 grade (American Society of Anesthesiology),
* and inability to comply with the follow-up protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8006 (Actual)
Dates: Start 1999-01; Primary Completion 2004-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure was the prevalence of recurrent goiter, incidental thyroid cancer and need for revision thyroid surgery. | folow-up at yearly intervals following thyroidectomy

SECONDARY OUTCOMES:
Secondary outcome measure was the postoperative morbidity rate (hypoparathyroidism, recurrent laryngeal nerve injury and bleeding). | 12-month follow-up after thyroidectomy

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Barczynski, MD, PhD, Principal Investigator — Jagiellonian University
Locations (1):
- Jagiellonian Univerity, Medical College, 3rd Department of general Surgery, Krakow, Malopolska, Poland

REFERENCES:
- [Background] Snook KL, Stalberg PL, Sidhu SB, Sywak MS, Edhouse P, Delbridge L. Recurrence after total thyroidectomy for benign multinodular goiter. World J Surg. 2007 Mar;31(3):593-8; discussion 599-600. doi: 10.1007/s00268-006-0135-0. PMID 17308855
- [Background] Wheeler MH. Total thyroidectomy for benign thyroid disease. Lancet. 1998 May 23;351(9115):1526-7. doi: 10.1016/S0140-6736(05)61116-6. No abstract available. PMID 10326531
- [Background] Ozbas S, Kocak S, Aydintug S, Cakmak A, Demirkiran MA, Wishart GC. Comparison of the complications of subtotal, near total and total thyroidectomy in the surgical management of multinodular goitre. Endocr J. 2005 Apr;52(2):199-205. doi: 10.1507/endocrj.52.199. PMID 15863948
- [Background] Moalem J, Suh I, Duh QY. Treatment and prevention of recurrence of multinodular goiter: an evidence-based review of the literature. World J Surg. 2008 Jul;32(7):1301-12. doi: 10.1007/s00268-008-9477-0. PMID 18305998
- [Background] Tezelman S, Borucu I, Senyurek Giles Y, Tunca F, Terzioglu T. The change in surgical practice from subtotal to near-total or total thyroidectomy in the treatment of patients with benign multinodular goiter. World J Surg. 2009 Mar;33(3):400-5. doi: 10.1007/s00268-008-9808-1. PMID 18958517
- [Background] Agarwal G, Aggarwal V. Is total thyroidectomy the surgical procedure of choice for benign multinodular goiter? An evidence-based review. World J Surg. 2008 Jul;32(7):1313-24. doi: 10.1007/s00268-008-9579-8. PMID 18449595
- [Background] Phitayakorn R, McHenry CR. Follow-up after surgery for benign nodular thyroid disease: evidence-based approach. World J Surg. 2008 Jul;32(7):1374-84. doi: 10.1007/s00268-008-9487-y. PMID 18311576
- [Background] Barczynski M, Konturek A, Cichon S. Randomized clinical trial of visualization versus neuromonitoring of recurrent laryngeal nerves during thyroidectomy. Br J Surg. 2009 Mar;96(3):240-6. doi: 10.1002/bjs.6417. PMID 19177420
- [Derived] Barczynski M, Konturek A, Stopa M, Cichon S, Richter P, Nowak W. Total thyroidectomy for benign thyroid disease: is it really worthwhile? Ann Surg. 2011 Nov;254(5):724-29; discussion 729-30. doi: 10.1097/SLA.0b013e3182360118. PMID 22005150